CLINICAL TRIAL: NCT00582881
Title: Immune Response to Small Nuclear Ribonucleoprotein Autoantigens
Brief Title: Characteristics and Disease Progression of Mixed Connective Tissue Disease and Systemic Lupus Erythematosus
Status: Recruiting | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Eric L. Greidinger, Associate Professor of Medicine, University of Miami
Other Study IDs: 20030724; 5R01AR043308-16 (NIH); 5R01AR043308-14 (NIH)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Mixed Connective Tissue Disease (MCTD); Systemic Lupus Erythematosus (SLE)
Keywords: Anti-RNP/Sm Autoantibody-Positive; MCTD; SLE
MeSH Terms: conditions — Mixed Connective Tissue Disease; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, cells, DNA, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Systemic lupus erythematosus (SLE) and mixed connective tissue disease (MCTD) are long-term autoimmune diseases in which the immune system attacks parts of the body. The abnormal immune reaction causes inflammation of and damage to various body parts and can affect joints, skin, kidneys, heart, lungs, blood vessels, and the brain. SLE and MCTD often affect young women, especially black and Hispanic women, and there is no known cure. Knowing more about SLE and MCTD will help in developing new and effective treatments. The purpose of this study is to characterize immune system abnormalities, genetic components, and disease progression in people with SLE and MCTD.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is an autoimmune disease in which the immune system produces antibodies against the body's healthy cells and tissues. These antibodies, called autoantibodies, contribute to the inflammation of various parts of the body and can cause damage to organs and tissues. Mixed connective tissue disease (MCTD) is another autoimmune disease that overlaps in terms of signs and symptoms with three other connective tissue diseases, including SLE. In both SLE and MCTD, the immune system appears to be abnormally activated by small nuclear ribonucleoprotein (snRNP) autoantigens. Furthermore, lung tissue, in particular, appears to be affected by the immune response induced by snRNP autoantigens. The causes of SLE and MCTD remain unknown. However, it is likely that a combination of genetic, environmental, and possibly hormonal factors work together to cause the diseases. Past studies suggest that several different genes may be involved in determining a person's likelihood of developing SLE or MCTD, which tissues and organs are affected, and the severity of the disease. The purpose of this study is to characterize immune system abnormalities, genetic components, and disease progression in people with SLE and MCTD.

Participants will attend up to four study visits, at intervals of at least 3 months, over the course of this study. Each study visit will include questionnaires, a physical exam, and possibly blood and/or urine collection. At the end of the study period, participants may choose to continue or discontinue participation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known rheumatic diseases including systemic lupus erythematosus, rheumatoid arthritis, connective tissue disease, undifferentiated connective tissue disease

Exclusion Criteria:

* Poor venous access, unstable medical problems or significant cardiopulmonary disease, anemia, leukopenia, thrombocytopenia, anticoagulation therapy, recent significant changes in medication or pregnacy. Patient cannot be taking large dose of corticosteroids (above 30mg per day) or cytotoxic drugs (cyclophosphamide, azathiprine, cyclosporine, methotrexate).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), mixed connective tissue disease (MCTD) or undifferentiated connective tissue disease (UCTD)
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2007-10 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Data characterizing immune cell responses and corresponding clinical data | Up to 4 visits at intervals of at least 3 months.
Phenotype measurement to include disease activity, disease severity, and functional status | up to 4 visits at intervals of at least 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric L. Greidinger, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No